CLINICAL TRIAL: NCT00837889
Title: Cognitive Impairment and Prognosis in Patients With Decompensated Heart Failure
Brief Title: Cognitive Impairment in Patients With Heart Failure
Acronym: CogImpairHF
Status: Completed | Type: Observational
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Sponsor
Other Study IDs: 164/08
Record Dates: First submitted 2009-02-03; First posted 2009-02-06 (Estimated); Last update posted 2025-08-11 (Actual); Status verified 2010-11

CONDITIONS: Heart Failure; Cognitive Impairment
Keywords: cognition; decompensation; heart failure; recompensation
MeSH Terms: conditions — Heart Failure; Cognitive Dysfunction | interventions — Diuretics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- decompensated heart failure patients
  Interventions: Drug: diuretics, inotropica
- chronic heart failure patients
- healthy controls

INTERVENTIONS:
Drug: diuretics, inotropica
  Groups: decompensated heart failure patients

SUMMARY:
The aim of the present study is threefold: investigating 1) specific cognitive impairments in patients with congestive heart failure, 2) whether cognitive impairments in patients with decompensated heart failure improve after medical recompensation and 3) whether cognitive functioning is related to the long-term prognosis (mortality, rehospitalisation) of those patients.

DETAILED DESCRIPTION:
The daily routine in clinical settings often shows cognitive impairments in patients with congestive heart failure. Recent studies reported declines in cognitive functioning such as executive functions, episodic memory, perceptual speed and attention. However, less is known regarding the differential impairments of cognitive functioning in patients with decompensated heart failure.

Study objectives:

1. Identifying specific cognitive impairments in patients with congestive heart failure compared to healthy controls
2. Evaluating the influence of acute decompensation in congestive heart failure on cognitive functioning
3. Investigating the effects of medical treatment on cognitive functioning in patients with decompensated heart failure
4. Exploring long-term effects of cognitive and physiological status on hospitalisation and/or mortality

Study design:

Cognitive functions of patients with decompensated heart (NYHA III-IV) failure are compared to age and gender matched patients with congestive heart failure (NYHA III-IV) without symptoms of cardiac decompensation and with healthy controls. Decompensated patients are tested before and after medical recompensation. For matched patients and controls, the pretest-posttest timing is based on the recompensation time of the respective patient with decompensated heart failure.

The neuropsychological test battery includes measures of episodic memory, working memory, short-term memory, executive functions, perceptual speed and intelligence. In addition, the study applied standardized questionnaires of self assessed quality of life and depression. Relevant physiological data, such as left ventricular systolic function and N-terminal pro brain natriuretic peptide (NT-pro-BNP), are recorded.

ELIGIBILITY:
Criteria of decompensated heart failure patients

Inclusion Criteria:

* decompensated heart failure patients
* NYHA III-IV
* ejection fraction < 35%

Exclusion Criteria:

* psychosis
* dementia
* major depression
* reanimation (<3month)
* patients with assist device system

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: university hospital, saarland
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-01; Primary Completion 2010-11 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
cognitive function in decompensated heart failure patients measured by a cognitive test battery | within 48h of hospitalisation
cognitive function before and after medical recompensation measured by a cognitive test battery | individual time to recompensate
differences in cognitive performance between decompensated heart failure patients, patients with chronic heart failure and healthy controls | 14 months (+/-2 month)

SECONDARY OUTCOMES:
all cause mortality | 12 month
long-term development of cognitive functioning in patients with heart failure after acute decompensation | 3, 6, 12 and 18 months after acute decompensation

CONTACTS AND LOCATIONS:
Overall Officials: Michael Böhm, MD, Principal Investigator — University Hospital, Saarland; Ingrid Kindermann, MD, Principal Investigator — University Hospital, Saarland; Denise Fischer, Psychologist, Principal Investigator — University Hospital, Saarland
Locations (2):
- Germany (2):
  - Department of Cardiology, University of the Saarland, Homburg, Saarland
  - Developmental Psychology Unit, Saarland University, Saarbrücken, Saarland

REFERENCES:
- [Background] Kindermann I, Fischer D, Karbach J, Link A, Walenta K, Barth C, Ukena C, Mahfoud F, Kollner V, Kindermann M, Bohm M. Cognitive function in patients with decompensated heart failure: the Cognitive Impairment in Heart Failure (CogImpair-HF) study. Eur J Heart Fail. 2012 Apr;14(4):404-13. doi: 10.1093/eurjhf/hfs015. PMID 22431406